CLINICAL TRIAL: NCT00710528
Title: A Phase 1 Sequential Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of CAL-101 in Patients With Select, Relapsed or Refractory Hematologic Malignancies
Brief Title: Dose Escalation Study of CAL-101 in Select Relapsed or Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Langdon Miller, M.D., VP Clinical Research, Onoclogy, Gilead Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-02
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Lymphoma, Non-Hodgkin (NHL); Acute Myeloid Leukemia (AML); Multiple Myeloma (MM)
Keywords: CLL; NHL; AML; MM; Phosphatidylinositol 3-kinase
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Multiple Myeloma | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one arm (Experimental)
  Interventions: Drug: CAL-101

INTERVENTIONS:
Drug: CAL-101 — CAL-101 50, 100, 150, 200, 350 mg capsules BID for 28 days CAL-101 150, 300 mg QD for 28 days CAL-101 150 mg BID 3 weeks on 1 week off for 28 days

SUMMARY:
The purpose of this study is to determine the dose that can be safely given to see what effect it may have on your cancer and to determine how the drug is distributed in the body.

DETAILED DESCRIPTION:
A Phase 1, sequential dose escalation followed by cohort expansion study of CAL-101, an oral inhibitor of PI3K delta, in patients with relapsed or refractory CLL, select B-cell NHL and AML.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18.
2. Has relapsed or refractory disease as defined by the following:

   * CLL - refractory to or relapsed after at least 2 prior therapies, including fludarabine, alone or in combination. Patients should not be eligible for transplantation (patients who are candidates for transplantation and have declined transplantation are eligible for this study).
   * B-cell NHL - refractory to or relapsed after at least 1 prior chemotherapy regimen and having received rituximab as a single agent or in combination with other therapies.
   * AML - refractory to or relapsed after at least 1 cycle of induction chemotherapy. Patients over the age of 70 who are not appropriate candidates for chemotherapy are eligible for this study.
   * MM - refractory to or relapsed after at least 2 prior chemotherapy regimens, including bortezomib and thalidomide or lenalidomide (except if the drug is contraindicated in a patient then this requirement is waived).
3. Disease status requirement:

   * For CLL patients, symptomatic disease that mandate treatment.
   * For B-cell NHL patients, has measurable disease by CT scan.
   * For AML patients, has > 10% blasts in the bone marrow for refractory or relapsed disease and > 20% blasts in the bone marrow if no prior chemotherapy.
   * For MM patients, has measurable disease defined by at least 1 of the following 3 measurements: serum M-protein > or = to 1 g/dL, urine M-protein > or = to 200 mg/24 h, or serum free light chain (FLC) assay with involved FLC level > or = to 10 mg/dL provided serum FLC ratio is abnormal.
4. WHO performance status of ≤ 2.
5. For men and women of child-bearing potential, willing to use adequate contraception (i.e., latex condom, cervical cap, diaphragm, abstinence, etc.) for the entire duration of the study.
6. Is able to provide written informed consent.

Exclusion Criteria:

1. Had radiotherapy, radioimmunotherapy, biological therapy, chemotherapy, or treatment with an investigational product within 4-weeks prior to screening.
2. For CLL or NHL patients, had treatment with a short course of corticosteroids for symptom relief within 1-week prior to screening.
3. Had alemtuzumab therapy within 12-weeks prior to screening.
4. For AML patients, had treatment with hydroxyurea within 1-week prior to screening.
5. Is pregnant or nursing.
6. Has significant, ongoing co-morbid conditions which would preclude safe delivery of the study drug.
7. Has had a transplant with current active graft-versus-host-disease.
8. Has known active central nervous system involvement of the malignancy.
9. Has active, serious infection requiring systemic therapy. Patients may receive prophylactic antibiotics and antiviral therapy at the discretion of the treating physician.
10. Has significant renal or liver dysfunction.
11. Has severe thrombocytopenia requiring platelet transfusion support, unless the diagnosis is AML.
12. Has a positive test for human immunodeficiency virus (HIV) antibodies.
13. Has active hepatitis B or C. Patients with serologic evidence of prior exposure are eligible.
14. Has poorly controlled diabetes mellitus.
15. Has taken a medication that is a potent inhibitor or inducer of cytochrome P450 3A4 within 1-week prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of CAL-101 and determine the dose limiting toxicity in patients with hematologic malignancies. | 28 days

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic parameters, pharmacodynamic effects and clinical response rate following CAL-101 treatment in patients with hematologic malignancies. | 28 Days

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Stanford Cancer Center, Palo Alto, California
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Medical College of Cornell, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Kahl BS, Spurgeon SE, Furman RR, Flinn IW, Coutre SE, Brown JR, Benson DM, Byrd JC, Peterman S, Cho Y, Yu A, Godfrey WR, Wagner-Johnston ND. A phase 1 study of the PI3Kdelta inhibitor idelalisib in patients with relapsed/refractory mantle cell lymphoma (MCL). Blood. 2014 May 29;123(22):3398-405. doi: 10.1182/blood-2013-11-537555. Epub 2014 Mar 10. PMID 24615778
- [Derived] Brown JR, Byrd JC, Coutre SE, Benson DM, Flinn IW, Wagner-Johnston ND, Spurgeon SE, Kahl BS, Bello C, Webb HK, Johnson DM, Peterman S, Li D, Jahn TM, Lannutti BJ, Ulrich RG, Yu AS, Miller LL, Furman RR. Idelalisib, an inhibitor of phosphatidylinositol 3-kinase p110delta, for relapsed/refractory chronic lymphocytic leukemia. Blood. 2014 May 29;123(22):3390-7. doi: 10.1182/blood-2013-11-535047. Epub 2014 Mar 10. PMID 24615777
- [Derived] Flinn IW, Kahl BS, Leonard JP, Furman RR, Brown JR, Byrd JC, Wagner-Johnston ND, Coutre SE, Benson DM, Peterman S, Cho Y, Webb HK, Johnson DM, Yu AS, Ulrich RG, Godfrey WR, Miller LL, Spurgeon SE. Idelalisib, a selective inhibitor of phosphatidylinositol 3-kinase-delta, as therapy for previously treated indolent non-Hodgkin lymphoma. Blood. 2014 May 29;123(22):3406-13. doi: 10.1182/blood-2013-11-538546. Epub 2014 Mar 10. PMID 24615776
- [Derived] Stevenson FK, Krysov S, Davies AJ, Steele AJ, Packham G. B-cell receptor signaling in chronic lymphocytic leukemia. Blood. 2011 Oct 20;118(16):4313-20. doi: 10.1182/blood-2011-06-338855. Epub 2011 Aug 3. PMID 21816833